CLINICAL TRIAL: NCT04871997
Title: A Real-world Study: Efficacy and Safety of Anlotinib for Advanced Non-small Cell Lung Cancer
Brief Title: A Real-world Study: Efficacy and Safety of Anlotinib for Advanced Non-small Cell Lung Cancer(NSCLC)
Status: Completed | Type: Observational
Sponsor: Qian Chu (Other)
Responsible Party: Sponsor-Investigator, Qian Chu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: S1040
Record Dates: First submitted 2021-04-26; First posted 2021-05-04 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: NSCLC
Keywords: NSCLC; anlotinib; PFS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All registered data are collected from real clinical practice cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A real-world study: Efficacy and safety of Anlotinib for advanced non-small cell lung cancer：This study aims to observe and explore the efficacy and safety of anlotinib in patients with advanced non-small cell lung cancer in the real world, and to summarize the treatment experience of a broad population.

DETAILED DESCRIPTION:
A real-world study: Efficacy and safety of Anlotinib for advanced non-small cell lung cancer：This study aims to observe and explore the efficacy and safety of anlotinib in patients with advanced non-small cell lung cancer in the real world, and to summarize the treatment experience of a broad population.This study is a non-interventional, prospective, observational, real-world case study and all registered data are collected from real clinical practice cases. Adult patients diagnosed as advanced non-small cell lung cancer and treated with anlotinib were included. At least one tumor lesion has not been subjected to local treatment such as irradiation in the past, and can be accurately measured, the longest diameter is ≥10 mm.The primary endpoint was progression-free survival (PFS) and the secondary endpoints included overall survival (OS), objective response rate (ORR), disease control rate (DCR) and safety.If the last patient reaches the main evaluation index or has intolerable toxic reaction, the observation will be finished, and the first one will prevail.Through Electronic Data Capture System (EDC) system, electronic case report form (eCRF) is used to replace paper-based case report form to collect and manage clinical trial data.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, no gender limit.
2. Diagnosed as advanced non-small cell lung cancer.
3. At least one tumor lesion has not been subjected to local treatment such as irradiation in the past, and can be accurately measured, the longest diameter is ≥10 mm.
4. Doctors evaluate the benefits of receiving Anlotinib treatment.
5. The patient voluntarily joins the project and signs the informed consent. If any of the above items is "No", the patient is not suitable for this study.

Exclusion Criteria:

1. Those who have been confirmed to be allergic to anlotinib and/or its excipients.
2. Patients with anlotinib contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed as advanced non-small cell lung cancer and treated with anlotinib were included，with no gender restriction
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2019.7-2022.7
  the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
overall survival (OS) | 2019.7-2022.7
  the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
objective response rate (ORR) | 2019.7-2022.7
  the percentage of patients on whom a therapy has some defined effect; for example, the cancer shrinks or disappears after treatment
disease control rate (DCR) | 2019.7-2022.7
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Chu, Principal Investigator — Tongji Hospital; Tienan Yi, Principal Investigator — Xiangyang Central Hospital; Youhong Dong, Principal Investigator — Xiangyang No.1 People's Hospital; Ruizhi Ran, Principal Investigator — The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture; Yang Fu, Principal Investigator — Xiangyang Hospital of Traditional Chinese Medicine; Guangqiao Qu, Principal Investigator — The Central Hospital of Xiao Gan; Jun Li, Principal Investigator — The Central Hospital of Xiao Gan; Yinping Li, Principal Investigator — The Central Hospital of Xiao Gan; Yanhua Xu, Principal Investigator — Jingzhou Central Hospital; Xinhua Xu, Principal Investigator — Yichang Central People's Hospital; Zhiguo Luo, Principal Investigator — Affiliated Taihe Hospital of Hubei University of Medicine; Fengjun Cao, Principal Investigator — Shiyan Renmin Hospital; Li Kuang, Principal Investigator — Dongfeng Hospital Affiliated to Hubei Medical College; Yifa Yin, Principal Investigator — Yichang Second People's Hospital; Guiming Chen, Principal Investigator — JingMen NO.2 People's Hospital
Locations (1):
- Hubei province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided